CLINICAL TRIAL: NCT01861080
Title: Observational Study of Clinical Characteristics and Prognostic Factors of Korean Hypertensives
Brief Title: Korean Registry of Target Organ Damages in Hypertension
Acronym: KorHR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dongtan Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Suk Won Choi, Kyu-Hyung Ryu, M.D., Professor, Dongtan Sacred Heart Hospital
Other Study IDs: 2012-005
Record Dates: First submitted 2013-05-16; First posted 2013-05-23 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Hypertension
Keywords: target organ damage; incident hypertension; cohort
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- incident hypertensives: Inclusion Criteria:
  * age≧30years
  * primary incident hypertension
  * signed informed consent

SUMMARY:
The objective of this study is to know prevalence of clinical or subclinical target organ damages in Korea hypertensives by constructing nationwide hypertension registry. We will register 5000 consecutive patients with incident hypertension at 20 major university hospitals in South Korea. We will investigate clinical/subclinical target organ damages, renin/aldosterone level and cardiovascular events in each patient.

DETAILED DESCRIPTION:
Background: the exact prevalence of target organ damages in Korean hypertensives are unknown.

Study Objective: to investigate the prevalence of target organ damages in Korean patients with incident hypertension.

Study Design: prospective, multi-center and observational study

Study Populaton: approximately 5000 consecutive patients with incident hypertension, who visited outpatients clinics and agreed to participate in the registry

Primary outcome

* Subclinical organ damages

  1. left ventricular hypertrophy on electrocardiogram or echocardiography
  2. increased intima media thickness of carotid artery (> 0.9 mm) or plaque
  3. increased pulse wave velocity (> 12 m/s)
  4. low estimated glomerular filtration rate (< 60 ml/min/1.73 m2) or creatinine clearance (<60 ml/min)
* Established CV or renal disease

  1. cerebrovascular disease: ischemic stroke; cerebral stroke; transient ischemic attack
  2. Heart disease: myocardial infarction; angina; coronary revascularization; heart failure
  3. Renal disease: diabetic retinopathy; serum creatinine M > 133, W > 124 mmol/L; proteinuria > 300 mg/24 hr
  4. Peripheral artery disease
  5. Advanced retinopathy: hemorrhage or exudates, papilledema

ELIGIBILITY:
Inclusion Criteria:

* age≧30years
* primary incident hypertension
* singed informed consent

Exclusion Criteria:

* participated in other clinical trials

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean patients with incident hypertensive, who visited university hospital
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2013-05; Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
left ventricular hypertrophy | at enrollment
  left ventricular hypertrophy on electrocardiogram or echocardiography Sokolow-Lyon > 38 mm; left ventricular mass index male >= 125 g/m2, female >=110 g/m2)
Intima media thickness of carotid artery | at enrollment
  increased intima media thickness of carotid artery (> 0.9 mm) or presence of plaque
pulse wave velocity | at enrollment
  increased pulse wave velocity (> 12 m/s)
kidney function | at enrollment
  low estimated glomerular filtration rate (< 60 ml/min/1.73 m2) or creatinine clearance (< 60 ml/min)
cerebrovascular accident | at enrollment
  ischemic stroke, cerebral hemorrhage, or transient ischemic attack confirmed by a neurologist
renal disease | at enrollment
  serum creatinine male > 1.5 mg/dl, female > 1.4 mg/dl; proteinuria > 300 mg/24hr
peripheral artery disease | at enrollment
  ankle to brachial blood pressure ratio < 0.9
retinopathy | at enrollment
  retinal hemorrhage or exudate, papilledema confirmed by an ophthalmologist

SECONDARY OUTCOMES:
Hypertension | at enrollment
  high blood pressure confirmed by ambulatory blood pressure monitoring (24hr average systolic blood pressure >=135 mm Hg, diastolic blood pressure >= 85 mm Hg
Dyslipidemia | at enrollment
  total cholesterol 190 mg/dl or LDL > 115 mg/dl, HDL male < 40 mg/dl, female < 46 mg/dl or triglyceride > 150 mg/dl
abnormal fasting plasma glucose | at enrollment
  abnormal fasting plasma glucose (102-125 mg/dl)
abdominal obesity | at enrollment
  waist circumference male > 102 cm, female > 88 cm
diabetes mellitus | at enrollment
  fasting plasma glucose >= 126 mg/dl; postload plasma glucose > 198 mg/dl

OTHER OUTCOMES:
major cardiovascular events | after follow-up period of 36 months
  death, stroke, myocardial infarction and heart failure(confirmed by a cardiologist)

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Hyung Ryu, MD, PhD, Principal Investigator — Dongtan Sacred Heart Hospital, Hallym University
Locations (1):
- Hallym University Dongtan Sacred Heart Hospital,, Hwaseong, Gyeonggido, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Choi SW, Han SW, Ok JS, Yoo BS, Shin MS, Park SH, Ryu KH. A multicenter cohort study of primary hypertension in Korea: study design and interim analysis of the Korean registry of target organ damage in hypertension (KorHR). Clin Hypertens. 2017 Aug 2;23:16. doi: 10.1186/s40885-017-0072-2. eCollection 2017. PMID 28794898